CLINICAL TRIAL: NCT01783366
Title: Nasogastric Tube Insertion Using Cook Airway Exchange Catheter in Anesthetized Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Collaborators: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Hyeon-Jeong Lee, ASSISTANT PROFESSOR, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNU03-2013-002; PNUYH03-2013-002 (Other: PUSAN NATIONAL UNIVERSITY YANGSAN HOSPITAL)
Record Dates: First submitted 2013-01-24; First posted 2013-02-04 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Elective Surgery of Gastrointestinal Tract; 100 Adults Aged Between 20 and 70 Years Old; ASA Physical Status of I or II
Keywords: nasogastric tube, tube exchange catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTROL (No Intervention): In the control group (Group A) inserting the lubricated NG tube through the nostril, at that time head maintained in the neutral position.
- tube-exchanger (Active Comparator): The tube-exchanger group (Group B) made use of tube-exchanger G36402 (CAEC, [cook medical, Bloomington, IN]) as a stylet that was lubricated and inserted within 20-F NGT until the tip of the tube-exchanger was at the tip of the NGT
  Interventions: Device: TUBE EXCHANGER

INTERVENTIONS:
Device: TUBE EXCHANGER
  Other Names: TUBE EXCHANGER USAGE
  Arms: tube-exchanger

SUMMARY:
we first examined whether use of tube exchange catheter during NGT insertion could increase the success rate on the first attempt of NGT insertion compared with conventional technique. We then addressed the question of whether the use of tube exchange catheter might decrease the possible occurrence of complication associated with YOON insertion.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status of I or II who were scheduled to undergo elective surgery of gastrointestinal tract with NGT insertion under general anesthesia were enrolled

Exclusion Criteria:

* Patients with maxillofacial trauma, inability to adequately protect airway, and esophageal abnormalities were excluded. Pregnant patients were also excluded from the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Number of attempt of NGT insertion | after successful insertion of NGT, within 1 hr
  After anesthetic induction, in the control group inserting the lubricated NG tube through the nostril, at that time head maintained in the neutral position. The tube-exchanger group made use of tube-exchanger as stylet within 20-F NGT. Success of appropriate NGT insertion through the nostrils until 70cm of NGT was considered with gurgling sounds on the auscultation over the epigastrium when 10ml of air was injected through the NGT and gastric contents aspiration via NGT. Total number of attempts until successful NGT insertion was recorded and tried at least three times, and was considered to have failed.
  Thus, procedure time would be the dependent factor of primary endpoin which could increse the success rate of NGT.
Procedure time of NGT insertion | after successful insertion of NGT, within 1 hr
  After anesthetic induction, in the control group inserting the lubricated NG tube through the nostril, at that time head maintained in the neutral position. The tube-exchanger group made use of tube-exchanger as stylet within 20-F NGT. Success of appropriate NGT insertion was considered with gurgling sounds on the auscultation over the epigastrium when 10ml of air was injected through the NGT and gastric contents aspiration via NGT. NGT insertion time recorded when the NGT begun to insert gently through the nostrils until 70cm of NGT.

SECONDARY OUTCOMES:
presence of bleeding of the larynx, and knotting or kinking of NGT under laryngoscopic view | after successful insertion of NGT within the time of completion of surgery, expected average within 6 hours
  The investigators examined the occurrence of complication associated with NGT insertion. After successful NGT insertion, we recorded presence of bleeding of the larynx, and knotting or kinking of NGT using laryngoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Pnuyh Anesthesia, Yangsan, South Korea